CLINICAL TRIAL: NCT04282395
Title: Improving Health Outcomes in African Americans With Type 2 Diabetes: A Culturally Tailored, Resilience-Based Diabetes Self-Management Education (RB-DSME) Intervention
Brief Title: Resilience-Based Diabetes Self-Management Education (RB-DSME) for African Americans
Acronym: TXSTRIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Mary Steinhardt, Principal Investigator (MPI), University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DK123146 (NIH)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes self-management; Church setting; African Americans; Health disparities; Resilience
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The primary goal of the project is to test the efficacy of a resilience-based diabetes self-management education intervention (RB-DSME) using a longitudinal, randomized control group design. Thirty-two AA churches are randomly assigned to the RB-DSME experimental group or a standard diabetes self-management education (DSME) control group, run in 8 cohorts over a 5-year period. Each cohort includes 4 churches (2 intervention, 2 control) with 10 participants in each group, run concurrently. Experimental and control groups participate in 8 weekly 1.5-hour classes, followed by 8 bimonthly (every other week) 1.5-hour support group sessions, followed by 2 every other month 1.5-hour booster sessions. Data are collected at baseline and also at 6 and 12 months post study entry; the specific diabetes-related outcomes are also measured at 24 months.
  During the in-person pause in research due to the pandemic, the intervention groups are held via Zoom and will continue in that format.
Who Masked: Participant, Care Provider
Masking Description: All study participants receive a behavioral intervention that is aimed at managing their diabetes condition, either a standard diabetes self-management education intervention or the experimental resilience-based diabetes self-management education intervention. Due to the nature of behavioral interventions, we are only able to mask the participants, care providers, and dietary recall outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience-Based Diabetes Self-Management Education (Experimental): The RB-DSME structure involves 8 weekly classes, 8 bimonthly support group sessions, and 2 booster sessions. The RB-DSME builds on foundational resilience resources (e.g., self-efficacy, social support), infusing novel resilience resources (e.g., adaptation to stress, finding positive meaning, spiritual coping) into the RB-DSME curriculum.
  Interventions: Behavioral: Resilience-Based Diabetes Self-Management Education
- Standard Diabetes Self-Management Education (Active Comparator): The scope and sequence of the standard diabetes self-management education (DSME) curriculum are aligned with national standards of the American Diabetes Association. DSME groups receive a 10-month intervention: 8 weekly educational sessions, followed by 8 bimonthly support group sessions, followed by 2 booster sessions.
  Interventions: Behavioral: Standard Diabetes Self-Management Education

INTERVENTIONS:
Behavioral: Resilience-Based Diabetes Self-Management Education — During the group sessions led by professional nurses, participants are provided information and group activities to enable them to more effectively manage their personal diabetes challenges. During the support group sessions, participants discuss personal challenges and solutions to diabetes self-management, using a more informal approach. Booster sessions are held to refresh participants' understanding of how resilience resources can sustain self-management behaviors and maintain improved T2DM health outcomes. The RB-DSME also incorporates cultural characteristics and preferences of African Americans (AAs), to include:
  * the location in community-based church settings,
  * recognition of cultural dietary preferences, and
  * emphasis on cultural/historical significance of resilience in AAs.
  Other Names: RB-DSME
  Arms: Resilience-Based Diabetes Self-Management Education
Behavioral: Standard Diabetes Self-Management Education — Control group sessions, led by professional nurses, cover topics such as:
  * causes and symptoms of type 2 diabetes,
  * glucose self-monitoring,
  * models for and principles of healthy eating, grocery shopping and dining out,
  * physical activity,
  * diabetes medications,
  * managing sick days and stress, and
  * community resources.
  Other Names: DSME
  Arms: Standard Diabetes Self-Management Education

SUMMARY:
African Americans are twice as likely to have type 2 diabetes as non-Hispanic Whites and are less likely to engage in effective diabetes self-management. There is a critical need for intensive lifestyle interventions that address the distress inherent in having the disease and the unique stressors faced by African Americans that may worsen diabetes-related health outcomes. Our program, Resilience-Based Diabetes Self-Management Education and Support, integrates resilience resources with diabetes self-management skills to enable African-American patients to manage the daily demands of the disease and improve long-term adherence to healthy lifestyle choices, thereby reducing the negative health burden of diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) costs the U.S. $327 billion annually, representing a 26% increase from 2012 to 2017. African Americans (AAs) are twice as likely to have T2DM as non-Hispanic Whites, have worse health outcomes, and are less likely to engage in self-management behaviors. Interventions addressing these disparities are urgently needed. Among AAs, T2DM-associated stress is often compounded by general life stress, which further constrains diabetes self-management and is associated with poor glucose control (A1C) and complications such as depression. The impact of stress on diabetes self-management and health outcomes may be attenuated by resilience: a resolve to succeed despite adversities. Even with evidence supporting resilience resources benefiting other health outcomes, there is a dearth of evidence-based T2DM resilience interventions. Building on our promising pilot work, this study uses our culturally tailored, theory-derived Resilience-Based Diabetes Self-Management Education (RB-DSME) intervention to help participants manage the psychosocial and behavioral demands of the disease. The study is designed as a 24-month, 2-arm, cluster randomized clinical trial and involves assigning AA churches to the RB-DSME or a standard DSME condition. Both groups receive a 10-month intervention: 8 weekly educational sessions, followed by 8 bimonthly support group sessions, followed by 2 booster sessions. To investigate the efficacy of RB-DSME, we compare RB-DSME to DSME on T2DM physical and mental health outcomes. To inform more targeted future interventions, we examine indirect effects of RB-DSME (vs DSME) on resilience resources, such as stress and coping. We also examine indirect effects of resilience resources on T2DM health outcomes through self-management behaviors, such as diet and exercise.

The specific aims of the study are:

Aim 1: To compare T2DM physical health outcomes (primary outcome: A1C) and T2DM mental health outcomes (primary outcome: depressive symptoms) in the RB-DSME group vs DSME group at 6, 12, and 24 months.

H1: Compared with DSME, RB-DSME will have improved T2DM physical health outcomes.

H2: Compared with DSME, RB-DSME will have improved T2DM mental health outcomes.

Aim 2: To test indirect effects of RB-DSME (vs DSME) on T2DM physical and mental health outcomes via resilience resources, self-management behaviors, and HPA axis function.

H3: RB-DSME (vs DSME) will improve resilience resources at 6 and 12 months, which will improve T2DM physical and mental health outcomes at 12 and 24 months.

H4: RB-DSME (vs DSME) driven improvements in resilience resources at 6 months will improve self-management and HPA axis function at 12 months, which will improve T2DM outcomes at 24 months.

The project will provide crucial guidance for addressing the T2DM burden among AAs by establishing the efficacy of the RB-DSME and identifying behavioral and biological mechanisms by which the program affects T2DM health outcomes. The long-term goal is to enable AAs to effectively manage T2DM and thus avoid its serious consequences, via RB-DSME interventions in a range of community settings.

ELIGIBILITY:
Inclusion Criteria: Participants must:

* be African American;
* be diagnosed with T2DM;
* be 18 years of age or older;
* have an A1C of 6.5 or higher; and
* not be currently participating in another T2DM management program.

Exclusion Criteria: Individuals will be excluded if they:

* are pregnant/lactating;
* have medical conditions for which changes in diet and/or physical activity would be contraindicated (e.g., hospitalization for heart disease during the past 6 months, diagnosed heart failure, kidney failure, or peripheral vascular disease requiring special diets and/or restricted physical activity severe enough to preclude walking three times per week, or active tuberculosis); or
* use glucocorticoid containing medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2025-04-26 (Estimated); Study Completion 2025-04-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin (A1C) at 6 months | Baseline and 6 months
  Glycosylated hemoglobin (A1C) provides a 3-month average of blood glucose levels and is used to determine changes in blood glucose levels over time. A blood sample is obtained through finger prick capillary blood collection and measured using the A1C Now Self Check (PTS Diagnostics, Indianapolis, IN). The A1C Now Self Check is a commercially available kit designed for home use and requires a finger prick similar to testing blood glucose with a handheld glucometer. The kit is a National Glycohemoglobin Standardization Program certified test that provides results in 5 minutes.
Change from baseline in glycosylated hemoglobin (A1C) at 12 months | Baseline and 12 months
  Glycosylated hemoglobin (A1C) provides a 3-month average of blood glucose levels and is used to determine changes in blood glucose levels over time. A blood sample is obtained through finger prick capillary blood collection and measured using the A1C Now Self Check (PTS Diagnostics, Indianapolis, IN). The A1C Now Self Check is a commercially available kit designed for home use and requires a finger prick similar to testing blood glucose with a handheld glucometer. The kit is a National Glycohemoglobin Standardization Program certified test that provides results in 5 minutes.
Change from baseline in glycosylated hemoglobin (A1C) at 24 months | Baseline and 24 months
  Glycosylated hemoglobin (A1C) provides a 3-month average of blood glucose levels and is used to determine changes in blood glucose levels over time. A blood sample is obtained through finger prick capillary blood collection and measured using the A1C Now Self Check (PTS Diagnostics, Indianapolis, IN). The A1C Now Self Check is a commercially available kit designed for home use and requires a finger prick similar to testing blood glucose with a handheld glucometer. The kit is a National Glycohemoglobin Standardization Program certified test that provides results in 5 minutes.
Change from baseline in depressive symptoms at 6 months | Baseline and 6 months
  The primary mental health outcome, Depressive Symptoms, is measured with the Patient Health Questionnaire-9 (PHQ-9; Cronbach's alpha reliability = .86), which measures the frequency and severity of depressive symptoms. The scale contains 9 items, each of which is rated on a 0-3 scale; higher scores indicate higher levels of depression.
Change from baseline in depressive symptoms at 12 months | Baseline and 12 months
  The primary mental health outcome, Depressive Symptoms, is measured with the Patient Health Questionnaire-9 (PHQ-9; Cronbach's alpha reliability = .86), which measures the frequency and severity of depressive symptoms. The scale contains 9 items, each of which is rated on a 0-3 scale; higher scores indicate higher levels of depression.
Change from baseline in depressive symptoms at 24 months | Baseline and 24 months
  The primary mental health outcome, Depressive Symptoms, is measured with the Patient Health Questionnaire-9 (PHQ-9; Cronbach's alpha reliability = .86), which measures the frequency and severity of depressive symptoms. The scale contains 9 items, each of which is rated on a 0-3 scale; higher scores indicate higher levels of depression.

SECONDARY OUTCOMES:
Change from baseline in dietary intake at 6 months | Baseline and 6 months
  Dietary intake is measured by trained interviewers who collect two 24-hour dietary recalls using the multiple pass technique by telephone (ensuring data for 1 weekend and 1 weekday) within 10 days of each data collection session (baseline, 6, 12 months). All recall data will be analyzed using the Nutrition Data System for Research (NDS-R; 2012, University of Minnesota). The NDS-R calculates key dietary variables including energy, macronutrients, total and added sugar, fiber, glycemic index, food/beverages servings/day, and a Healthy Eating Index (HEI).
Change from baseline in dietary intake at 12 months | Baseline and 12 months
  Dietary intake is measured by trained interviewers who collect two 24-hour dietary recalls using the multiple pass technique by telephone (ensuring data for 1 weekend and 1 weekday) within 10 days of each data collection session (baseline, 6, 12 months). All recall data will be analyzed using the Nutrition Data System for Research (NDS-R; 2012, University of Minnesota). The NDS-R calculates key dietary variables including energy, macronutrients, total and added sugar, fiber, glycemic index, food/beverages servings/day, and a Healthy Eating Index (HEI).
Change from baseline in physical activity at 6 months | Baseline and 6 months
  Physical activity is measured with accelerometers (wGT3X-BT, Actigraph LLC, Pensacola, FL). Physical activity is measured for 7 days in the same week as the in-person data collection session and the dietary recalls (baseline, 6, 12 months). All accelerometer data are immediately downloaded and wear time assessed. If the participant does not have at least 4 days with ≥8 hours of wear time, the accelerometer is re-issued to the participant. The following data from all acceptable days are available: minutes and percent time spent in light physical activity, moderate to vigorous physical activity, and sedentary behavior. Adult cutoffs are used to quantify and classify accelerometry data.
Change from baseline in physical activity at 12 months | Baseline and 12 months
  Physical activity is measured with accelerometers (wGT3X-BT, Actigraph LLC, Pensacola, FL). Physical activity is measured for 7 days in the same week as the in-person data collection session and the dietary recalls (baseline, 6, 12 months). All accelerometer data are immediately downloaded and wear time assessed. If the participant does not have at least 4 days with ≥8 hours of wear time, the accelerometer is re-issued to the participant. The following data from all acceptable days are available: minutes and percent time spent in light physical activity, moderate to vigorous physical activity, and sedentary behavior. Adult cutoffs are used to quantify and classify accelerometry data.
Change from baseline in diabetes self-care at 6 months | Baseline and 6 months
  Diabetes self-care is measured by the 12-item Self-Care Inventory-Revised (SCI-R), which assesses perceived diabetes self-care adherence. The SCI-R is designed on a 1 to 5 Likert-type scale from 1 (never do it) to 5 (always do this). Total possible scores range from 12 to 60, with higher scores indicating enhanced diabetes self-care. The Cronbach's alpha reliability = .87.
Change from baseline in diabetes self-care at 12 months | Baseline and 12 months
  Diabetes self-care is measured by the 12-item Self-Care Inventory-Revised (SCI-R), which assesses perceived diabetes self-care adherence. The SCI-R is designed on a 1 to 5 Likert-type scale from 1 (never do it) to 5 (always do this). Total possible scores range from 12 to 60, with higher scores indicating enhanced diabetes self-care. The Cronbach's alpha reliability = .87.
Change from baseline in physiological stress (HPA axis function) at 6 months | Baseline and 6 months
  Hair cortisol and DHEA are assessed by collecting proximal 3 cm of scalp-near hair. Once all hair samples are collected for each cohort, they are shipped to and analyzed. Steroid levels are determined using a commercial high sensitivity enzyme-linked immunoassay kit (Salimetrics LLC, State College, PA), per manufacturer's protocol. A professional hair stylist collects the samples to ease any participant concerns.
  During the in-person research pause due to the pandemic, hair cortisol will be conducted via self-administered protocol by participants at their home. The hair sample collected will be identical in size to the one collected in person.
Change from baseline in physiological stress (HPA axis function) at 12 months | Baseline and 12 months
  Hair cortisol and DHEA are assessed by collecting proximal 3 cm of scalp-near hair. Once all hair samples are collected for each cohort, they are shipped to and analyzed. Steroid levels are determined using a commercial high sensitivity enzyme-linked immunoassay kit (Salimetrics LLC, State College, PA), per manufacturer's protocol. A professional hair stylist collects the samples to ease any participant concerns.
Change from baseline in fasting blood glucose levels at 6 months | Baseline and 6 months
  Fasting plasma concentrations of glucose is determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA).
Change from baseline in fasting blood glucose levels at 12 months | Baseline and 12 months
  Fasting plasma concentrations of glucose is determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA).
Change from baseline in fasting blood glucose levels at 24 months | Baseline and 24 months
  Fasting plasma concentrations of glucose is determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA).
Change from baseline in cholesterol levels at 6 months | Baseline and 6 months
  Cholesterol (including total, LDL, and HDL) is determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA)
Change from baseline in cholesterol levels at 12 months | Baseline and 12 months
  Cholesterol (including total, LDL, and HDL) is determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA)
Change from baseline in cholesterol levels at 24 months | Baseline and 24 months
  Cholesterol (including total, LDL, and HDL) is determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA)
Change from baseline in triglycerides at 6 months | Baseline and 6 months
  Fasting plasma concentrations of triglycerides are determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA).
Change from baseline in triglycerides at 12 months | Baseline and 12 months
  Fasting plasma concentrations of triglycerides are determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA).
Change from baseline in triglycerides at 24 months | Baseline and 24 months
  Fasting plasma concentrations of triglycerides are determined through finger prick capillary blood collection and analyzed enzymatically with Alere reagent on a Cholestech LDX analyzer (Alere, Waltham, MA).
Change from baseline in body mass index (BMI) at 6 months | Baseline and 6 months
  Body mass index (BMI) is measured with the following formula: BMI = (weight in kg)/(height in m)2. For the calculation, body weight is measured using a Tanita Professional Digital Scale (Model BF350). Participants wear street clothes and no shoes; coats and belts are removed. Height is determined using a portable stadiometer, Seca 214.
Change from baseline in body mass index (BMI) at 12 months | Baseline and 12 months
  Body mass index (BMI) is measured with the following formula: BMI = (weight in kg)/(height in m)2. For the calculation, body weight is measured using a Tanita Professional Digital Scale (Model BF350). Participants wear street clothes and no shoes; coats and belts are removed. Height is determined using a portable stadiometer, Seca 214.
Change from baseline in body mass index (BMI) at 24 months | Baseline and 24 months
  Body mass index (BMI) is measured with the following formula: BMI = (weight in kg)/(height in m)2. For the calculation, body weight is measured using a Tanita Professional Digital Scale (Model BF350). Participants wear street clothes and no shoes; coats and belts are removed. Height is determined using a portable stadiometer, Seca 214.
Change from baseline in waist circumference at 6 months | Baseline and 6 months
  Waist circumference is measured to the nearest 0.1 cm using a non-stretchable standard tape measure attached to a spring balance, 0.1 cm above the iliac crest on a horizontal plane.
Change from baseline in waist circumference at 12 months | Baseline and 12 months
  Waist circumference is measured to the nearest 0.1 cm using a non-stretchable standard tape measure attached to a spring balance, 0.1 cm above the iliac crest on a horizontal plane.
Change from baseline in waist circumference at 24 months | Baseline and 24 months
  Waist circumference is measured to the nearest 0.1 cm using a non-stretchable standard tape measure attached to a spring balance, 0.1 cm above the iliac crest on a horizontal plane.
Change from baseline in blood pressure at 6 months | Baseline and 6 months
  Blood pressure (systolic and diastolic) is measured with an Omron HEM-907XL Automatic Inflation Blood Pressure Monitor (Omron, Philadelphia, PA). Following a 5-minute rest period, the monitor takes 3 consecutive readings 1 minute apart and displays the average, following American Heart Association guidelines.
Change from baseline in blood pressure at 12 months | Baseline and 12 months
  Blood pressure (systolic and diastolic) is measured with an Omron HEM-907XL Automatic Inflation Blood Pressure Monitor (Omron, Philadelphia, PA). Following a 5-minute rest period, the monitor takes 3 consecutive readings 1 minute apart and displays the average, following American Heart Association guidelines.
Change from baseline in blood pressure at 24 months | Baseline and 24 months
  Blood pressure (systolic and diastolic) is measured with an Omron HEM-907XL Automatic Inflation Blood Pressure Monitor (Omron, Philadelphia, PA). Following a 5-minute rest period, the monitor takes 3 consecutive readings 1 minute apart and displays the average, following American Heart Association guidelines.
Change from baseline in diabetes distress at 6 months | Baseline and 6 months
  Diabetes distress is measured with the 4-item Diabetes Distress Scale (Cronbach's alpha reliability = .90), assessing the emotional burden due to having T2DM. Each item is rated from 1 (not a problem) to 6 (serious problem). Total possible scores range from 4 to 24, with higher scores indicating more distress with the burden of diabetes.
Change from baseline in diabetes distress at 12 months | Baseline and 12 months
  Diabetes distress is measured with the 4-item Diabetes Distress Scale (Cronbach's alpha reliability = .90), assessing the emotional burden due to having T2DM. Each item is rated from 1 (not a problem) to 6 (serious problem). Total possible scores range from 4 to 24, with higher scores indicating more distress with the burden of diabetes.
Change from baseline in diabetes distress at 24 months | Baseline and 24 months
  Diabetes distress is measured with the 4-item Diabetes Distress Scale (Cronbach's alpha reliability = .90), assessing the emotional burden due to having T2DM. Each item is rated from 1 (not a problem) to 6 (serious problem). Total possible scores range from 4 to 24, with higher scores indicating more distress with the burden of diabetes.
Change from baseline in general perceived stress at 6 months | Baseline and 6 months
  General stress is assessed with the 10-item Perceived Stress Scale (Cronbach's alpha reliability = .82), which measures the degree to which situations in one's life are appraised as stressful. Each item is rated on a 0 (never) to 4 (very often) scale. Total possible scores range from 0 to 40, with higher scores indicating higher levels of general stress.
Change from baseline in general perceived stress at 12 months | Baseline and 12 months
  General stress is assessed with the 10-item Perceived Stress Scale (Cronbach's alpha reliability = .82), which measures the degree to which situations in one's life are appraised as stressful. Each item is rated on a 0 (never) to 4 (very often) scale. Total possible scores range from 0 to 40, with higher scores indicating higher levels of general stress.
Change from baseline in general perceived stress at 24 months | Baseline and 24 months
  General stress is assessed with the 10-item Perceived Stress Scale (Cronbach's alpha reliability = .82), which measures the degree to which situations in one's life are appraised as stressful. Each item is rated on a 0 (never) to 4 (very often) scale. Total possible scores range from 0 to 40, with higher scores indicating higher levels of general stress.
Change from baseline in sleep quantity and quality at 6 months | Baseline and 6 months
  Sleep quantity and quality are measured with a sleep scale involving 9 items, designed as a Likert-type scale with each item measured on a 0 (not during the past month) to 3 (3 times during the past month). Eight items measure sleep problems and one item is a sleep quality rating (0=very good to 3=very bad). Total possible points range from 0 to 27, with higher scores indicating more sleep problems and poorer sleep quality.
Change from baseline in sleep quantity and quality at 12 months | Baseline and 12 months
  Sleep quantity and quality are measured with a sleep scale involving 9 items, designed as a Likert-type scale with each item measured on a 0 (not during the past month) to 3 (3 times during the past month). Eight items measure sleep problems and one item is a sleep quality rating (0=very good to 3=very bad). Total possible points range from 0 to 27, with higher scores indicating more sleep problems and poorer sleep quality.
Change from baseline in spiritual coping at 6 months | Baseline and 6 months
  Spiritual coping is measured with the Spiritual-Centered Coping subscale of the Africultural Coping Systems Inventory. Spiritual coping behaviors are grounded in the participant's perceived connection with the Creator or the Universe. The Likert-type contains 8 items, each ranging from 0 (did not use) to 3 (used a great deal). Total possible scores range from 0 to 24, with higher scores indicating higher levels of spiritual coping. Cronbach alpha reliability = .79.
Change from baseline in spiritual coping at 12 months | Baseline and 12 months
  Spiritual coping is measured with the Spiritual-Centered Coping subscale of the Africultural Coping Systems Inventory. Spiritual coping behaviors are grounded in the participant's perceived connection with the Creator or the Universe. The Likert-type contains 8 items, each ranging from 0 (did not use) to 3 (used a great deal). Total possible scores range from 0 to 24, with higher scores indicating higher levels of spiritual coping. Cronbach alpha reliability = .79.
Change from baseline in self-efficacy at 6 months | Baseline and 6 months
  Self-efficacy is measured with the Modified Generalized Self-Efficacy Scale, which measures how confident individuals are in managing their diabetes, despite life's stressors. The scale contains 10 Likert-type items rated from 0 (not true at all) to 4 (true nearly all of the time). Total scores range from 0 to 40, with higher scores indicating higher self-efficacy (Cronbach's alpha reliability = .76 - .90).
Change from baseline in self-efficacy at 12 months | Baseline and 12 months
  Self-efficacy is measured with the Modified Generalized Self-Efficacy Scale, which measures how confident individuals are in managing their diabetes, despite life's stressors. The scale contains 10 Likert-type items rated from 0 (not true at all) to 4 (true nearly all of the time). Total scores range from 0 to 40, with higher scores indicating higher self-efficacy (Cronbach's alpha reliability = .76 - .90).
Change from baseline in finding positive meaning at 6 months | Baseline and 6 months
  The Positive Meaning Scale is used to measure the extent to which individuals find positive meaning in the context of having a diagnosis of type 2 diabetes. The scale contains 5 Likert-type items rated from 0 (definitely no) to 3 (definitely yes). Total scores range from 0 to 15, with higher scores indicating higher levels of finding positive meaning (Cronbach's alpha reliability = .73).
Change from baseline in finding positive meaning at 12 months | Baseline and 12 months
  The Positive Meaning Scale is used to measure the extent to which individuals find positive meaning in the context of having a diagnosis of type 2 diabetes. The scale contains 5 Likert-type items rated from 0 (definitely no) to 3 (definitely yes). Total scores range from 0 to 15, with higher scores indicating higher levels of finding positive meaning (Cronbach's alpha reliability = .73).
Change from baseline in adaptive coping strategies at 6 months | Baseline and 6 months
  The Coping Orientations to Problems Experienced Scale (14 adaptive coping items) is used to measure cognitive and behavioral strategies that enable an individual to handle adversity. The scale is a Likert-type scale in which participants rate on a 0 (I haven't been doing this AT ALL) to 3 (I've been doing this A LOT) scale. Total scores range from 0 to 42, with higher scores indicating higher levels of adaptive coping (Cronbach's alpha reliability = .73 - .79).
Change from baseline in adaptive coping strategies at 12 months | Baseline and 12 months
  The Coping Orientations to Problems Experienced Scale (14 adaptive coping items) is used to measure cognitive and behavioral strategies that enable an individual to handle adversity. The scale is a Likert-type scale in which participants rate on a 0 (I haven't been doing this AT ALL) to 3 (I've been doing this A LOT) scale. Total scores range from 0 to 42, with higher scores indicating higher levels of adaptive coping (Cronbach's alpha reliability = .73 - .79).
Change from baseline in adaptation to stress at 6 months | Baseline and 6 months
  The Connor-Davidson Resilience Scale is used to identify personal qualities that enable an individual to persevere and adapt positively in the face of adversity. The scale is a Likert-type instrument that contains 10 items, each of which is rated on a 1 (not at all true) to 4 (exactly true) scale. Total scores range from 10 to 40, with higher scores indicating higher levels of adaptation to stress (Cronbach's alpha reliability = .85). For confirmatory purposes, we also use the Brief Resilience Scale contains 6 items that also assess adaptation to stress, with a rating scale of 1 (strongly disagree) to 5 (strongly agree).
Change from baseline in adaptation to stress at 12 months | Baseline and 12 months
  The Connor-Davidson Resilience Scale is used to identify personal qualities that enable an individual to persevere and adapt positively in the face of adversity. The scale is a Likert-type instrument that contains 10 items, each of which is rated on a 1 (not at all true) to 4 (exactly true) scale. Total scores range from 10 to 40, with higher scores indicating higher levels of adaptation to stress (Cronbach's alpha reliability = .85). For confirmatory purposes, we also use the Brief Resilience Scale contains 6 items that also assess adaptation to stress, with a rating scale of 1 (strongly disagree) to 5 (strongly agree).
Change from baseline in coping with discrimination at 6 months | Baseline and 6 months
  The Coping with Discrimination Scale is used to determine how minority individuals respond to discrimination. We use 22 Likert-type items from the original 25-item scale, each of which is rated from 1 (never like me) to 6 (always like me). Total scores range from 22 - 132; higher scores indicate higher levels of coping. Scale reliability (Cronbach's alpha) ranges from .73 - .90.
Change from baseline in coping with discrimination at 12 months | Baseline and 12 months
  The Coping with Discrimination Scale is used to determine how minority individuals respond to discrimination. We use 22 Likert-type items from the original 25-item scale, each of which is rated from 1 (never like me) to 6 (always like me). Total scores range from 22 - 132; higher scores indicate higher levels of coping. Scale reliability (Cronbach's alpha) ranges from .73 - .90.
Change from baseline in emotional regulation at 6 months | Baseline and 6 months
  The Brief Version of the Emotional Regulation Scale (DERS-16) is used to measure awareness and acceptance of emotions, as well as strategies used to regulate emotions. The scale consists of 16 Likert-type items with possible responses to each item ranging from 1 (almost never) to 5 (almost always). Total possible scores range from 16 to 80, with higher scores indicating less effective strategies used to regulate emotions. Scale reliability (Cronbach's alpha) ranges from 0.85 to 0.88.
Change from baseline in emotional regulation at 12 months | Baseline and 12 months
  The Brief Version of the Emotional Regulation Scale (DERS-16) is used to measure awareness and acceptance of emotions, as well as strategies used to regulate emotions. The scale consists of 16 Likert-type items with possible responses to each item ranging from 1 (almost never) to 5 (almost always). Total possible scores range from 16 to 80, with higher scores indicating less effective strategies used to regulate emotions. Scale reliability (Cronbach's alpha) ranges from 0.85 to 0.88.
Change from baseline in social support at 6 months | Baseline and 6 months
  The Multi-Dimensional Scale of Perceived Social Support is used to measure an individual's perceived adequacy of support for diabetes self-management from family, friends, and significant others. The instrument consists of 12 Likert-type items and each item is rated on a 1 (very strongly disagree) to 7 (very strongly agree) scale. Total possible scores range from 12 to 84, with higher scores indicating higher levels of perceived social support. Scale reliability (Cronbach's alpha) ranges from .84 to .92.
Change from baseline in social support at 12 months | Baseline and 12 months
  The Multi-Dimensional Scale of Perceived Social Support is used to measure an individual's perceived adequacy of support for diabetes self-management from family, friends, and significant others. The instrument consists of 12 Likert-type items and each item is rated on a 1 (very strongly disagree) to 7 (very strongly agree) scale. Total possible scores range from 12 to 84, with higher scores indicating higher levels of perceived social support. Scale reliability (Cronbach's alpha) ranges from .84 to .92.

CONTACTS AND LOCATIONS:
Overall Officials: Mary A. Steinhardt, EdD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woo J, Lehrer HM, Tabibi D, Cebulske L, Tanaka H, Steinhardt M. The Association of Multidimensional Sleep Health With HbA1c and Depressive Symptoms in African American Adults With Type 2 Diabetes. Psychosom Med. 2024 May 1;86(4):307-314. doi: 10.1097/PSY.0000000000001298. PMID 38724038